CLINICAL TRIAL: NCT03984578
Title: Window of Opportunity Study With Neoadjuvant Pembrolizumab in Colorectal Cancer
Brief Title: Window of Opportunity Study in Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WoOCRC
Record Dates: First submitted 2019-06-04; First posted 2019-06-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab; Capecitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Newly Diagnosed Colon cancers (Experimental): Pre-operative CAPEOX 1 cycle Pre-operative Pembrolizumab 2 cycles with cycle 1 on Day 1 (concurrent with start of CAPEOX) and cycle 2 on Day 22.
  Interventions: Drug: CAPEOX; Drug: Pembrolizumab; Procedure: Surgical resection
- Newly Diagnosed Rectal Cancers (Experimental): Following completion of neo-adjuvant chemo-radiotherapy, 2 cycles of pre-operative Pembrolizumab administered 3 weeks apart.
  Interventions: Drug: Capecitabine/ 5-FU; Drug: Pembrolizumab; Procedure: Surgical resection
- Newly Diagnosed Colon and Rectal Cancers Referred for Pre-Operative Chemotherapy (Experimental): Neoadjuvant pembrolizumab 3-weekly for a maximum of 6 doses to be administered along with XELOX chemotherapy, and additional 1 dose pembrolizumab.
  Interventions: Drug: CAPEOX/Pembrolizumab; Drug: Pembrolizumab alone; Procedure: Surgical resection

INTERVENTIONS:
Drug: CAPEOX — Oral Capecitabine: 1000mg/m2 twice a day from Day 1 to 14 of a 3-week cycle, and IV Oxaliplatin: 130mg/m2 on Day 1
  Arms: Newly Diagnosed Colon cancers
Drug: Pembrolizumab — IV infusion of 200mg on Day 1 and Day 22
  Other Names: Keytruda
  Arms: Newly Diagnosed Colon cancers
Drug: Capecitabine/ 5-FU — Capecitabine: Oral dose of 825mg/m2/day twice a day on radiation days with concurrent radiation median 50.4 Gy/ 28 fractions; or 5-FU: 225mg/m2/day concurrent with radiation
  Arms: Newly Diagnosed Rectal Cancers
Drug: Pembrolizumab — IV infusion of 200mg on Day 1 of each cycle
  Other Names: Keytruda
  Arms: Newly Diagnosed Rectal Cancers
Drug: CAPEOX/Pembrolizumab — * Oral Capecitabine: 1000mg/m2 twice a day from Day 1 to 14 of a 3-week cycle.
  * IV Oxaliplatin: 130mg/m2 on Day 1 of a 3-week cycle.
  * Pembrolizumab: IV infusion of 200mg on Day 1 of a 3-week cycle.
  Arms: Newly Diagnosed Colon and Rectal Cancers Referred for Pre-Operative Chemotherapy
Drug: Pembrolizumab alone — IV infusion of 200mg 21 days from the last CAPEOX/Pembrolizumab combination dose.
  Other Names: Keytruda
  Arms: Newly Diagnosed Colon and Rectal Cancers Referred for Pre-Operative Chemotherapy
Procedure: Surgical resection — Performed after all medical intervention.

SUMMARY:
This is a window of opportunity translational study investigating the use of pre-operative pembrolizumab and chemotherapy or chemoradiotherapy in non-metastatic colorectal cancer.

DETAILED DESCRIPTION:
Patients with radiologically-assessed locally advanced non-metastatic colorectal cancer will receive the following treatment before surgery:

Newly Diagnosed Colon cancers:

One cycle of CAPEOX chemotherapy Two cycles of Pembrolizumab on Day 1 (concurrent with CAPEOX chemotherapy) and Day 22.

Newly Diagnosed Rectal cancers:

Following completion of chemo-radiotherapy with 5-fluorouracil (5-FU)/ capecitabine, patients will receive 2 cycles of Pembrolizumab given 3 weeks apart.

Colon and Rectal Cancer Patients Referred for Pre-Operative Chemotherapy:

Neoadjuvant pembrolizumab 200 mg 3-weekly for a maximum of 6 doses to be administered along with XELOX chemotherapy and additional 1 dose pembrolizumab 200 mg followed by standard of care (SOC) tumour resection.

Pre-operative biopsy and surgical samples as well as blood will be collected for translational studies.

ELIGIBILITY:
Inclusion Criteria:

1. For patients with colon cancer (Group 1): Adenocarcinoma of the colon (radiologic T4 and/or N2) OR rectal adenocarcinoma with positive lymph nodes and/or threatened/positive circumferential resection margin (CRM).

   Radiological staging is based on the degree of tumor infiltration beyond the serosa:
   * rT1-2 tumors - no tumor extension beyond the serosa.
   * rT3 tumors - tumor extension <5 mm beyond the serosa.
   * rT4 tumors - tumor extension ≥5 mm beyond the serosa.

   Lymph nodes are considered positive if they are more than 10 mm in short axis diameter or demonstrate an irregular contour:
   * rN0 - absence of nodal involvement.
   * rN1 - involvement of 1-3 nodes.
   * rN2 - involvement of ≥ 4 nodes.
2. For patients with rectal cancer (Group 1): Patients with rectal adenocarcinoma must have completed neoadjuvant chemoradiation therapy (or planned to receive neoadjuvant chemoradiation at point of recruitment).
3. Colon or Rectal Cancer patients referred for preoperative chemotherapy (Group 2).

   Note: Patients may be included at any point during the preoperative chemotherapy phase and have pembrolizumab administered concurrently with the remaining cycles of preoperative chemotherapy.
4. Male/female participants who are at least 21 years of age on the day of signing informed consent with histologically confirmed diagnosis of colorectal adenocarcinoma.
5. Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: a) Not a woman of childbearing potential (WOCBP) OR b) A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
6. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
7. Tumor evaluated to have sufficient tissue for translational studies
8. Have provided sufficient archival tumor tissue sample.
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation/randomization.
10. Have adequate organ function as defined in the following table. Specimens must be collected within 14 days prior to the start of study treatment.

    Adequate Organ Function Laboratory:
    * Absolute neutrophil count (ANC): ≥1500/μL.
    * Platelets: ≥100 000/μL.
    * Hemoglobin: ≥9.0 g/dL or ≥5.6 mmol/L.
    * Creatinine OR Measured or calculated creatinine clearance: ≤1.5 × Upper Limit of Normal (ULN) OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
    * Total bilirubin: ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN.
    * Alanine Aminotransferase and Aspartate Aminotransferase: ≤2.5 × ULN.
    * Coagulation - International normalized ratio (INR) OR prothrombin time (PT) OR Activated partial thromboplastin time (aPTT): ≤1.5 × ULN.
11. Are not on current anti-HCV treatment for subjects with chronic infection by HCV. For subjects who have had anti-HCV therapy, the last dose of anti-HCV medication should be at least 4 weeks before first dose of pembrolizumab.

    Note: Screening for chronic HCV infection will be done if subject's HCV status is not already known.
12. Have HBV viral load under 100 IU/mL with or without treatment, for subjects with chronic hepatitis B infection.

    * HBV viral load must be less than 100 IU/mL on at least 4 weeks of anti-viral therapy prior to first dose of pembrolizumab. Subjects on active HBV therapy with viral loads under 100 IU/mL should stay on the same therapy throughout study treatment. Subjects who are anti-HBc (+), negative for HBs Ag, negative for anti-HBs, and have an HBV viral load under 100 IU/mL do not require HBV anti-viral prophylaxis

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation of subject number. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has any sign of distant metastases or need for emergency surgery.
3. Has past history of bowel perforation and abdominal fistula, unless medically treated (e.g. by stoma) or deemed to still be suitable for pre-operative systemic therapy; a recent history of bowel resection (within past 12 months) and/or patients with radiological evidence of active bowel obstruction.
4. Has intercurrent illness, including but not limited to infections and unstable angina pectoris.
5. Is on anticoagulation therapy (warfarin, low molecular weight heparin, rivaroxaban).
6. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, and CD137).
7. Has received prior systemic anti-cancer therapy including investigational agents within 1 year prior to allocation, except capecitabine as neoadjuvant therapy for patients with rectal cancer.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

   Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
8. Has received prior radiotherapy within 1 year of start of study treatment or planned radiotherapy prior to surgery, except radiotherapy received as neoadjuvant therapy for patients with rectal cancer.
9. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
10. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device for cancer within 1 year prior to the first dose of study treatment.

    Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
11. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
12. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
13. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
16. Has an active infection requiring systemic therapy.
17. Has Human Immunodeficiency Virus (HIV).
18. Has a known history of active TB (Bacillus Tuberculosis).
19. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
22. Has dual active HBV infection [HBsAg (+) and/or detectable HBV DNA] and HCV infection [anti-HCV Ab (+) and detectable HCV RNA] at study entry.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Tumour immune gene expression signature | From time of first tumour biopsy before treatment to time of tumour resection performed 1-3 weeks after last dose of neoadjuvant treatment
  Gene expression of key immune genes will be assayed and immune gene expression scores such as IFN-gamma Gene Expression Profile (GEP) signature score (Ayers et al. 2017 JCI) will be compared before (biopsy) and after treatment (surgery).
Pathology regression | From time of first tumour biopsy before treatment to time of tumour resection performed 1-3 weeks after last dose of neoadjuvant treatment
  A change in viable tumour after treatment will be measured by pathologist using tumour regression grade and major pathologic regression.
Immune T-cell infiltration before and after treatment | From time of first tumour biopsy before treatment to time of tumour resection performed 1-3 weeks after last dose of neoadjuvant treatment
  The change in immune cell infiltration will be measured by pathologists through immunohistochemistry and/or immuno-fluorescence.

SECONDARY OUTCOMES:
Relative proportion/ percentage of the different immune cell states or immune cell types as inferred from single cell or bulk gene expression profiling | At time of tumour resection performed 1-3 weeks after last dose of neoadjuvant treatment
  Single cell RNA sequencing, bulk genomics & bulk transcriptomics will be used to describe the enrichment of different immune cell states or cell types
Relative distribution (percentage) of immune cells with specific expression of lineage markers | At time of tumour resection performed 1-3 weeks after last dose of neoadjuvant treatment
  Flow cytometry will be used to determine the proportions of immune cell types with specific lineage marker expression including CD45, CD4, CD8, PDL1 and LAG3
Percentage of cell viability and cell death at fixed time points (e.g. 24 or 48 hours) | At time of tumour resection performed 1-3 weeks after last dose of neoadjuvant treatment
  Functional assays of immune cell immunoreactivity will be used to determine the proportion of target cell kill of paired immune cell and target cell

CONTACTS AND LOCATIONS:
Overall Officials: Iain Tan, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (3):
- Singapore (3):
  - National Cancer Centre Singapore, Singapore
  - Singapore General Hospital, Singapore
  - Sengkang General Hospital, Singapore